CLINICAL TRIAL: NCT01459302
Title: Family Studies in Neuromuscular Disorders
Brief Title: Genetic Study of Familial and Sporadic ALS/Motor Neuron Disease, Miyoshi Myopathy and Other Neuromuscular Disorders
Status: Withdrawn | Type: Observational
Why Stopped: This study is not a clinical trial.
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Other Study IDs: H-13019
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Amyotrophic Lateral Sclerosis; Frontotemporal Dementia; PLS; Motor Neuron Disease; Lou Gehrigs Disease; Familial Disease; Amyotrophic Lateral Sclerosis, Sporadic; Muscular Dystrophy; Miyoshi Myopathy; Amyotrophic Lateral Sclerosis With Dementia
Keywords: FALS; ALS; SALS; MND; SOD1; ALS GENES; PLS; PMA; ALS/FTD; FAMILIAL ALS; SPORADIC ALS; GENETICS; FTD; Miyoshi myopathy
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Frontotemporal Dementia; Motor Neuron Disease; Amyotrophic lateral sclerosis 1; Muscular Dystrophies; Miyoshi myopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA(plus Serum, plasma, frozen cells when available) will be obtained from the initial blood or saliva sample for genetic study. RNA, skin cells or lymphoblast cells may be obtained and stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Familial and Sporadic ALS: Individuals with ALS and families with a history of two or more people in the family who have had ALS or other forms of motor neuron disease.

SUMMARY:
The investigators laboratory has been studying families with a history of ALS for more than 30 years and is continuing to use new ways to understand how genes may play a role in ALS, motor neuron disease and other neuromuscular disorders.

The purpose of this study is to identify additional genes that may cause or put a person at risk for either familial ALS (meaning 2 or more people in a family who have had ALS), sporadic ALS, or other forms of motor neuron disease in the hopes of improving diagnosis and treatment. As new genes are found that may be linked to ALS in families or individuals, the investigators can then further study how that gene may be contributing to the disease by studying it down to the protein and molecular level. This includes all forms of ALS, motor neuron disease and ALS with fronto-temporal dementia(ALS/FTD). We also continue to study other forms of neuromuscular disease such as Miyoshi myopathy, FSH dystrophy and other forms of muscular dystrophy by looking at the genes that may be associated with them.

There have been a number of genes identified that are associated with both familial and sporadic ALS, with the SOD1, C9orf72, and FUS genes explaining the majority of the cases. However, for about 25% of families with FALS, the gene(s) are still unknown.

The investigators also will continue to work with families already identified to carry one of the known genes associated with ALS.

DETAILED DESCRIPTION:
Participants will be asked to provide a blood sample ( or sometimes saliva or skin sample) and to complete a couple of questionnaires regarding their overall medical health. Medical records will need to be reviewed for all those diagnosed with one of the study diseases to allow the researchers to review details of their clinical disease symptoms, neurological exams and test results.

Participants do not need to travel to Massachusetts for this study. Samples can be obtained locally at no costs to the participant. Family members may be included in the study depending on family history and their relationship to the affected individual.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of or family history of ALS,MND,ALS with dementia, or PLS.
* diagnosis of Miyoshi myopathy
* willingness to provide a blood sample for study use

Exclusion Criteria:

* unwilling to provide a blood or saliva sample

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals diagnosed with ALS, motor neuron disease, PLS, ALS with dementia, Miyoshi Myopathy, some muscular dystrophies and spouse/population controls. Some family members may be eligible to participate as well.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
identification of new genes that may contribute to ALS | Up to 9 years
  identification and reporting of any new genes that may be associated with individuals or families with ALS is a primary goal to provide better diagnostics as well as new targets for treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Brown Jr., D Phil,MD, Principal Investigator — U Mass Medical School
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Background] Nicolas A, Kenna KP, Renton AE, Ticozzi N, Faghri F, Chia R, Dominov JA, Kenna BJ, Nalls MA, Keagle P, Rivera AM, van Rheenen W, Murphy NA, van Vugt JJFA, Geiger JT, Van der Spek RA, Pliner HA, Shankaracharya, Smith BN, Marangi G, Topp SD, Abramzon Y, Gkazi AS, Eicher JD, Kenna A; ITALSGEN Consortium; Mora G, Calvo A, Mazzini L, Riva N, Mandrioli J, Caponnetto C, Battistini S, Volanti P, La Bella V, Conforti FL, Borghero G, Messina S, Simone IL, Trojsi F, Salvi F, Logullo FO, D'Alfonso S, Corrado L, Capasso M, Ferrucci L; Genomic Translation for ALS Care (GTAC) Consortium; Moreno CAM, Kamalakaran S, Goldstein DB; ALS Sequencing Consortium; Gitler AD, Harris T, Myers RM; NYGC ALS Consortium; Phatnani H, Musunuri RL, Evani US, Abhyankar A, Zody MC; Answer ALS Foundation; Kaye J, Finkbeiner S, Wyman SK, LeNail A, Lima L, Fraenkel E, Svendsen CN, Thompson LM, Van Eyk JE, Berry JD, Miller TM, Kolb SJ, Cudkowicz M, Baxi E; Clinical Research in ALS and Related Disorders for Therapeutic Development (CReATe) Consortium; Benatar M, Taylor JP, Rampersaud E, Wu G, Wuu J; SLAGEN Consortium; Lauria G, Verde F, Fogh I, Tiloca C, Comi GP, Soraru G, Cereda C; French ALS Consortium; Corcia P, Laaksovirta H, Myllykangas L, Jansson L, Valori M, Ealing J, Hamdalla H, Rollinson S, Pickering-Brown S, Orrell RW, Sidle KC, Malaspina A, Hardy J, Singleton AB, Johnson JO, Arepalli S, Sapp PC, McKenna-Yasek D, Polak M, Asress S, Al-Sarraj S, King A, Troakes C, Vance C, de Belleroche J, Baas F, Ten Asbroek ALMA, Munoz-Blanco JL, Hernandez DG, Ding J, Gibbs JR, Scholz SW, Floeter MK, Campbell RH, Landi F, Bowser R, Pulst SM, Ravits JM, MacGowan DJL, Kirby J, Pioro EP, Pamphlett R, Broach J, Gerhard G, Dunckley TL, Brady CB, Kowall NW, Troncoso JC, Le Ber I, Mouzat K, Lumbroso S, Heiman-Patterson TD, Kamel F, Van Den Bosch L, Baloh RH, Strom TM, Meitinger T, Shatunov A, Van Eijk KR, de Carvalho M, Kooyman M, Middelkoop B, Moisse M, McLaughlin RL, Van Es MA, Weber M, Boylan KB, Van Blitterswijk M, Rademakers R, Morrison KE, Basak AN, Mora JS, Drory VE, Shaw PJ, Turner MR, Talbot K, Hardiman O, Williams KL, Fifita JA, Nicholson GA, Blair IP, Rouleau GA, Esteban-Perez J, Garcia-Redondo A, Al-Chalabi A; Project MinE ALS Sequencing Consortium; Rogaeva E, Zinman L, Ostrow LW, Maragakis NJ, Rothstein JD, Simmons Z, Cooper-Knock J, Brice A, Goutman SA, Feldman EL, Gibson SB, Taroni F, Ratti A, Gellera C, Van Damme P, Robberecht W, Fratta P, Sabatelli M, Lunetta C, Ludolph AC, Andersen PM, Weishaupt JH, Camu W, Trojanowski JQ, Van Deerlin VM, Brown RH Jr, van den Berg LH, Veldink JH, Harms MB, Glass JD, Stone DJ, Tienari P, Silani V, Chio A, Shaw CE, Traynor BJ, Landers JE. Genome-wide Analyses Identify KIF5A as a Novel ALS Gene. Neuron. 2018 Mar 21;97(6):1267-1288. doi: 10.1016/j.neuron.2018.02.027. PMID 29566793
- [Background] Cammack AJ, Atassi N, Hyman T, van den Berg LH, Harms M, Baloh RH, Brown RH, van Es MA, Veldink JH, de Vries BS, Rothstein JD, Drain C, Jockel-Balsarotti J, Malcolm A, Boodram S, Salter A, Wightman N, Yu H, Sherman AV, Esparza TJ, McKenna-Yasek D, Owegi MA, Douthwright C; Alzheimer's Disease Neuroimaging Initiative; McCampbell A, Ferguson T, Cruchaga C, Cudkowicz M, Miller TM. Prospective natural history study of C9orf72 ALS clinical characteristics and biomarkers. Neurology. 2019 Oct 22;93(17):e1605-e1617. doi: 10.1212/WNL.0000000000008359. Epub 2019 Oct 2. PMID 31578300
- [Background] de Majo M, Topp SD, Smith BN, Nishimura AL, Chen HJ, Gkazi AS, Miller J, Wong CH, Vance C, Baas F, Ten Asbroek ALMA, Kenna KP, Ticozzi N, Redondo AG, Esteban-Perez J, Tiloca C, Verde F, Duga S, Morrison KE, Shaw PJ, Kirby J, Turner MR, Talbot K, Hardiman O, Glass JD, de Belleroche J, Gellera C, Ratti A, Al-Chalabi A, Brown RH, Silani V, Landers JE, Shaw CE. ALS-associated missense and nonsense TBK1 mutations can both cause loss of kinase function. Neurobiol Aging. 2018 Nov;71:266.e1-266.e10. doi: 10.1016/j.neurobiolaging.2018.06.015. Epub 2018 Jun 25. PMID 30033073
- [Background] Smith BN, Topp SD, Fallini C, Shibata H, Chen HJ, Troakes C, King A, Ticozzi N, Kenna KP, Soragia-Gkazi A, Miller JW, Sato A, Dias DM, Jeon M, Vance C, Wong CH, de Majo M, Kattuah W, Mitchell JC, Scotter EL, Parkin NW, Sapp PC, Nolan M, Nestor PJ, Simpson M, Weale M, Lek M, Baas F, Vianney de Jong JM, Ten Asbroek ALMA, Redondo AG, Esteban-Perez J, Tiloca C, Verde F, Duga S, Leigh N, Pall H, Morrison KE, Al-Chalabi A, Shaw PJ, Kirby J, Turner MR, Talbot K, Hardiman O, Glass JD, De Belleroche J, Maki M, Moss SE, Miller C, Gellera C, Ratti A, Al-Sarraj S, Brown RH Jr, Silani V, Landers JE, Shaw CE. Mutations in the vesicular trafficking protein annexin A11 are associated with amyotrophic lateral sclerosis. Sci Transl Med. 2017 May 3;9(388):eaad9157. doi: 10.1126/scitranslmed.aad9157. PMID 28469040
- [Background] van Rheenen W, Shatunov A, Dekker AM, McLaughlin RL, Diekstra FP, Pulit SL, van der Spek RA, Vosa U, de Jong S, Robinson MR, Yang J, Fogh I, van Doormaal PT, Tazelaar GH, Koppers M, Blokhuis AM, Sproviero W, Jones AR, Kenna KP, van Eijk KR, Harschnitz O, Schellevis RD, Brands WJ, Medic J, Menelaou A, Vajda A, Ticozzi N, Lin K, Rogelj B, Vrabec K, Ravnik-Glavac M, Koritnik B, Zidar J, Leonardis L, Groselj LD, Millecamps S, Salachas F, Meininger V, de Carvalho M, Pinto S, Mora JS, Rojas-Garcia R, Polak M, Chandran S, Colville S, Swingler R, Morrison KE, Shaw PJ, Hardy J, Orrell RW, Pittman A, Sidle K, Fratta P, Malaspina A, Topp S, Petri S, Abdulla S, Drepper C, Sendtner M, Meyer T, Ophoff RA, Staats KA, Wiedau-Pazos M, Lomen-Hoerth C, Van Deerlin VM, Trojanowski JQ, Elman L, McCluskey L, Basak AN, Tunca C, Hamzeiy H, Parman Y, Meitinger T, Lichtner P, Radivojkov-Blagojevic M, Andres CR, Maurel C, Bensimon G, Landwehrmeyer B, Brice A, Payan CA, Saker-Delye S, Durr A, Wood NW, Tittmann L, Lieb W, Franke A, Rietschel M, Cichon S, Nothen MM, Amouyel P, Tzourio C, Dartigues JF, Uitterlinden AG, Rivadeneira F, Estrada K, Hofman A, Curtis C, Blauw HM, van der Kooi AJ, de Visser M, Goris A, Weber M, Shaw CE, Smith BN, Pansarasa O, Cereda C, Del Bo R, Comi GP, D'Alfonso S, Bertolin C, Soraru G, Mazzini L, Pensato V, Gellera C, Tiloca C, Ratti A, Calvo A, Moglia C, Brunetti M, Arcuti S, Capozzo R, Zecca C, Lunetta C, Penco S, Riva N, Padovani A, Filosto M, Muller B, Stuit RJ; PARALS Registry; SLALOM Group; SLAP Registry; FALS Sequencing Consortium; SLAGEN Consortium; NNIPPS Study Group; Blair I, Zhang K, McCann EP, Fifita JA, Nicholson GA, Rowe DB, Pamphlett R, Kiernan MC, Grosskreutz J, Witte OW, Ringer T, Prell T, Stubendorff B, Kurth I, Hubner CA, Leigh PN, Casale F, Chio A, Beghi E, Pupillo E, Tortelli R, Logroscino G, Powell J, Ludolph AC, Weishaupt JH, Robberecht W, Van Damme P, Franke L, Pers TH, Brown RH, Glass JD, Landers JE, Hardiman O, Andersen PM, Corcia P, Vourc'h P, Silani V, Wray NR, Visscher PM, de Bakker PI, van Es MA, Pasterkamp RJ, Lewis CM, Breen G, Al-Chalabi A, van den Berg LH, Veldink JH. Genome-wide association analyses identify new risk variants and the genetic architecture of amyotrophic lateral sclerosis. Nat Genet. 2016 Sep;48(9):1043-8. doi: 10.1038/ng.3622. Epub 2016 Jul 25. PMID 27455348
- [Background] Kenna KP, van Doormaal PT, Dekker AM, Ticozzi N, Kenna BJ, Diekstra FP, van Rheenen W, van Eijk KR, Jones AR, Keagle P, Shatunov A, Sproviero W, Smith BN, van Es MA, Topp SD, Kenna A, Miller JW, Fallini C, Tiloca C, McLaughlin RL, Vance C, Troakes C, Colombrita C, Mora G, Calvo A, Verde F, Al-Sarraj S, King A, Calini D, de Belleroche J, Baas F, van der Kooi AJ, de Visser M, Ten Asbroek AL, Sapp PC, McKenna-Yasek D, Polak M, Asress S, Munoz-Blanco JL, Strom TM, Meitinger T, Morrison KE; SLAGEN Consortium; Lauria G, Williams KL, Leigh PN, Nicholson GA, Blair IP, Leblond CS, Dion PA, Rouleau GA, Pall H, Shaw PJ, Turner MR, Talbot K, Taroni F, Boylan KB, Van Blitterswijk M, Rademakers R, Esteban-Perez J, Garcia-Redondo A, Van Damme P, Robberecht W, Chio A, Gellera C, Drepper C, Sendtner M, Ratti A, Glass JD, Mora JS, Basak NA, Hardiman O, Ludolph AC, Andersen PM, Weishaupt JH, Brown RH Jr, Al-Chalabi A, Silani V, Shaw CE, van den Berg LH, Veldink JH, Landers JE. NEK1 variants confer susceptibility to amyotrophic lateral sclerosis. Nat Genet. 2016 Sep;48(9):1037-42. doi: 10.1038/ng.3626. Epub 2016 Jul 25. PMID 27455347
- [Background] Fogh I, Lin K, Tiloca C, Rooney J, Gellera C, Diekstra FP, Ratti A, Shatunov A, van Es MA, Proitsi P, Jones A, Sproviero W, Chio A, McLaughlin RL, Soraru G, Corrado L, Stahl D, Del Bo R, Cereda C, Castellotti B, Glass JD, Newhouse S, Dobson R, Smith BN, Topp S, van Rheenen W, Meininger V, Melki J, Morrison KE, Shaw PJ, Leigh PN, Andersen PM, Comi GP, Ticozzi N, Mazzini L, D'Alfonso S, Traynor BJ, Van Damme P, Robberecht W, Brown RH, Landers JE, Hardiman O, Lewis CM, van den Berg LH, Shaw CE, Veldink JH, Silani V, Al-Chalabi A, Powell J. Association of a Locus in the CAMTA1 Gene With Survival in Patients With Sporadic Amyotrophic Lateral Sclerosis. JAMA Neurol. 2016 Jul 1;73(7):812-20. doi: 10.1001/jamaneurol.2016.1114. PMID 27244217
- [Background] Smith BN, Ticozzi N, Fallini C, Gkazi AS, Topp S, Kenna KP, Scotter EL, Kost J, Keagle P, Miller JW, Calini D, Vance C, Danielson EW, Troakes C, Tiloca C, Al-Sarraj S, Lewis EA, King A, Colombrita C, Pensato V, Castellotti B, de Belleroche J, Baas F, ten Asbroek AL, Sapp PC, McKenna-Yasek D, McLaughlin RL, Polak M, Asress S, Esteban-Perez J, Munoz-Blanco JL, Simpson M; SLAGEN Consortium; van Rheenen W, Diekstra FP, Lauria G, Duga S, Corti S, Cereda C, Corrado L, Soraru G, Morrison KE, Williams KL, Nicholson GA, Blair IP, Dion PA, Leblond CS, Rouleau GA, Hardiman O, Veldink JH, van den Berg LH, Al-Chalabi A, Pall H, Shaw PJ, Turner MR, Talbot K, Taroni F, Garcia-Redondo A, Wu Z, Glass JD, Gellera C, Ratti A, Brown RH Jr, Silani V, Shaw CE, Landers JE. Exome-wide rare variant analysis identifies TUBA4A mutations associated with familial ALS. Neuron. 2014 Oct 22;84(2):324-31. doi: 10.1016/j.neuron.2014.09.027. Epub 2014 Oct 22. PMID 25374358
- [Result] Kwiatkowski TJ Jr, Bosco DA, Leclerc AL, Tamrazian E, Vanderburg CR, Russ C, Davis A, Gilchrist J, Kasarskis EJ, Munsat T, Valdmanis P, Rouleau GA, Hosler BA, Cortelli P, de Jong PJ, Yoshinaga Y, Haines JL, Pericak-Vance MA, Yan J, Ticozzi N, Siddique T, McKenna-Yasek D, Sapp PC, Horvitz HR, Landers JE, Brown RH Jr. Mutations in the FUS/TLS gene on chromosome 16 cause familial amyotrophic lateral sclerosis. Science. 2009 Feb 27;323(5918):1205-8. doi: 10.1126/science.1166066. PMID 19251627
- [Result] Shatunov A, Mok K, Newhouse S, Weale ME, Smith B, Vance C, Johnson L, Veldink JH, van Es MA, van den Berg LH, Robberecht W, Van Damme P, Hardiman O, Farmer AE, Lewis CM, Butler AW, Abel O, Andersen PM, Fogh I, Silani V, Chio A, Traynor BJ, Melki J, Meininger V, Landers JE, McGuffin P, Glass JD, Pall H, Leigh PN, Hardy J, Brown RH Jr, Powell JF, Orrell RW, Morrison KE, Shaw PJ, Shaw CE, Al-Chalabi A. Chromosome 9p21 in sporadic amyotrophic lateral sclerosis in the UK and seven other countries: a genome-wide association study. Lancet Neurol. 2010 Oct;9(10):986-94. doi: 10.1016/S1474-4422(10)70197-6. PMID 20801717
- [Result] Blauw HM, Al-Chalabi A, Andersen PM, van Vught PW, Diekstra FP, van Es MA, Saris CG, Groen EJ, van Rheenen W, Koppers M, Van't Slot R, Strengman E, Estrada K, Rivadeneira F, Hofman A, Uitterlinden AG, Kiemeney LA, Vermeulen SH, Birve A, Waibel S, Meyer T, Cronin S, McLaughlin RL, Hardiman O, Sapp PC, Tobin MD, Wain LV, Tomik B, Slowik A, Lemmens R, Rujescu D, Schulte C, Gasser T, Brown RH Jr, Landers JE, Robberecht W, Ludolph AC, Ophoff RA, Veldink JH, van den Berg LH. A large genome scan for rare CNVs in amyotrophic lateral sclerosis. Hum Mol Genet. 2010 Oct 15;19(20):4091-9. doi: 10.1093/hmg/ddq323. Epub 2010 Aug 4. PMID 20685689
- [Result] Ticozzi N, LeClerc AL, Keagle PJ, Glass JD, Wills AM, van Blitterswijk M, Bosco DA, Rodriguez-Leyva I, Gellera C, Ratti A, Taroni F, McKenna-Yasek D, Sapp PC, Silani V, Furlong CE, Brown RH Jr, Landers JE. Paraoxonase gene mutations in amyotrophic lateral sclerosis. Ann Neurol. 2010 Jul;68(1):102-7. doi: 10.1002/ana.21993. PMID 20582942
- [Result] van Es MA, Veldink JH, Saris CG, Blauw HM, van Vught PW, Birve A, Lemmens R, Schelhaas HJ, Groen EJ, Huisman MH, van der Kooi AJ, de Visser M, Dahlberg C, Estrada K, Rivadeneira F, Hofman A, Zwarts MJ, van Doormaal PT, Rujescu D, Strengman E, Giegling I, Muglia P, Tomik B, Slowik A, Uitterlinden AG, Hendrich C, Waibel S, Meyer T, Ludolph AC, Glass JD, Purcell S, Cichon S, Nothen MM, Wichmann HE, Schreiber S, Vermeulen SH, Kiemeney LA, Wokke JH, Cronin S, McLaughlin RL, Hardiman O, Fumoto K, Pasterkamp RJ, Meininger V, Melki J, Leigh PN, Shaw CE, Landers JE, Al-Chalabi A, Brown RH Jr, Robberecht W, Andersen PM, Ophoff RA, van den Berg LH. Genome-wide association study identifies 19p13.3 (UNC13A) and 9p21.2 as susceptibility loci for sporadic amyotrophic lateral sclerosis. Nat Genet. 2009 Oct;41(10):1083-7. doi: 10.1038/ng.442. Epub 2009 Sep 6. PMID 19734901
- [Result] Wu CH, Fallini C, Ticozzi N, Keagle PJ, Sapp PC, Piotrowska K, Lowe P, Koppers M, McKenna-Yasek D, Baron DM, Kost JE, Gonzalez-Perez P, Fox AD, Adams J, Taroni F, Tiloca C, Leclerc AL, Chafe SC, Mangroo D, Moore MJ, Zitzewitz JA, Xu ZS, van den Berg LH, Glass JD, Siciliano G, Cirulli ET, Goldstein DB, Salachas F, Meininger V, Rossoll W, Ratti A, Gellera C, Bosco DA, Bassell GJ, Silani V, Drory VE, Brown RH Jr, Landers JE. Mutations in the profilin 1 gene cause familial amyotrophic lateral sclerosis. Nature. 2012 Aug 23;488(7412):499-503. doi: 10.1038/nature11280. PMID 22801503
- [Result] Gonzalez-Perez P, Cirulli ET, Drory VE, Dabby R, Nisipeanu P, Carasso RL, Sadeh M, Fox A, Festoff BW, Sapp PC, McKenna-Yasek D, Goldstein DB, Brown RH Jr, Blumen SC. Novel mutation in VCP gene causes atypical amyotrophic lateral sclerosis. Neurology. 2012 Nov 27;79(22):2201-8. doi: 10.1212/WNL.0b013e318275963b. Epub 2012 Nov 14. PMID 23152587
- [Result] Ticozzi N, Vance C, Leclerc AL, Keagle P, Glass JD, McKenna-Yasek D, Sapp PC, Silani V, Bosco DA, Shaw CE, Brown RH Jr, Landers JE. Mutational analysis reveals the FUS homolog TAF15 as a candidate gene for familial amyotrophic lateral sclerosis. Am J Med Genet B Neuropsychiatr Genet. 2011 Apr;156B(3):285-90. doi: 10.1002/ajmg.b.31158. Epub 2011 Jan 13. PMID 21438137